CLINICAL TRIAL: NCT06945900
Title: Emergency Medical Services (EMS) Telehealth to Speed STEMI Reperfusion (THOR)
Brief Title: Emergency Medical Services (EMS) Telehealth to Speed STEMI Reperfusion
Acronym: THOR
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Duke Endowment (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00094324
Record Dates: First submitted 2025-04-15; First posted 2025-04-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Heart Attack; Reperfusion therapy; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telehealth — Paramedics will utilize Telehealth for STEMI patients during transport to determine appropriate care steps.

SUMMARY:
The aim of this study is to evaluate the impact of a Telehealth program on the time from First Medical Contact (FMC) to Reperfusion in STEMI (ST-elevation myocardial infarction) patients, by supporting local paramedics in their care delivery.

DETAILED DESCRIPTION:
STEMI (ST-elevation myocardial infarction) is the most severe type of heart attack and carries a 30-day mortality of nearly 8%. Reperfusion therapy is the mainstay of treatment for STEMI, either by percutaneous coronary intervention (PCI) or fibrinolytics. Delays in reperfusion are associated with negative health outcomes. Specifically, each 30-minute delay in reperfusion corresponds to a 7.5% decrease in 1-year survival. The current body of literature clearly shows that rural EMS agencies often have longer transport times, which makes the 90-minute first medical contact (FMC) to PCI time goal difficult to achieve. Approximately 16% of Americans live more than an hour from a PCI-capable facility, reinforcing the need for timely therapies in rural prehospital settings to decrease heart muscle damage (disability) and mortality. An analysis of a large national EMS database, which showed that FMC to PCI times were longer for patients treated by rural EMS agencies even after these times were adjusted for distance to destination hospital.8In addition, preliminary data for Cherokee Tribal EMS, serving the Eastern Band of Cherokee Indians on the Qualla Boundary and its surrounding communities, show that none of their patients who called 9-1-1 for a STEMI received reperfusion within the AHA time goal. The American College of Cardiology and AHA support prehospital fibrinolytics when timely PCI cannot be performed. STEMI telehealth programs have yet to be implemented and tested in the United States.

ELIGIBILITY:
Inclusion Criteria:

* All patients calling 9-1-1 in Wilkes County with possible STEMI as determined by the on scene paramedics will be included in the data.

Exclusion Criteria:

* As this is a Quality Surveillance study, subjects will not be excluded.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients calling 9-1-1 in the Wilkes County that present with a possible STEMI as determined by the on scene paramedics.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
First Medical Contact to Reperfusion Time | Year 2
  FMC to reperfusion time will be recorded in a study database. Data will be aggregated from patients before (baseline) and after EMS telehealth STEMI program implementation. FMC to reperfusion time will be reported as a mean with standard deviation and as a median with interquartile range.
First Medical Contact to Electrocardiogram (EKG) time | Year 2
  FMC to EKG time will be recorded in a study database. Data will be aggregated from patients before (baseline) and after EMS telehealth STEMI program implementation. Time will be reported as a mean with standard deviation and as a median with interquartile range.
Electrocardiogram (EKG) to Activation time | Year 2
  FMC to activation time will be recorded in a study database. Data will be aggregated from patients before (baseline) and after EMS telehealth STEMI program implementation. Time will be reported as a mean with standard deviation and as a median with interquartile range.
Activation to reperfusion [by fibrinolytic or PCI] time) | Year 2
  Activation to reperfusion [by fibrinolytic or PCI] time) will be recorded in a study database. Data will be aggregated from patients before (baseline) and after EMS telehealth STEMI program implementation. Time will be reported as a mean with standard deviation and as a median with interquartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stopyra, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT06945900/Prot_000.pdf